CLINICAL TRIAL: NCT00142766
Title: Sedation Management in Pediatric Patients Supported on Mechanical Ventilation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Gustavus and Louise Pfeiffer Research Foundation (Other)
Responsible Party: Principal Investigator, Martha Curley, Ellen and Robert Kapito Professor in Nursing Science, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21HD045020 (NIH)
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Respiratory Failure
Keywords: Sedation; Mechanical ventilation; Critical illness; Analgesic; Opioid Withdrawal; Benzodiazepine Withdrawal; Nurse
MeSH Terms: conditions — Respiratory Insufficiency; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Nurse Implemented Goal-Directed Comfort Algorithm — See description

SUMMARY:
The purpose of this two-year project is to pilot test an intervention to change sedation management in pediatric patients supported on mechanical ventilation for acute respiratory failure in the pediatric intensive care unit (PICU). While ensuring patient comfort is an integral part of pediatric critical care, analgesic and sedative use in this patient population is associated with injury; specifically, comfort medications may depress spontaneous ventilation and prolong the duration of mechanical ventilation. Additionally, drug tolerance develops over time and may precipitate iatrogenic abstinence syndrome (chemical withdrawal) when the patient no longer requires sedation. Alternatively, suboptimal comfort management contributes to the patient not breathing synchronously with the ventilator and/or self-removal of breathing tubes.

Our group has developed and validated a nurse-implemented sedation algorithm (set of specific instructions) to guide titration of comfort medications that may optimize patient comfort and reduce the risk of under-medication, but this algorithm needs to be evaluated further. We hypothesize that pediatric patients managed per sedation protocol will experience fewer days of mechanical ventilation than patients receiving usual care. This research has the potential of revolutionizing sedation practices that are driven by and synchronized to patient needs.

DETAILED DESCRIPTION:
We propose a two-year project to pilot test and evaluate an intervention to change sedation management in pediatric patients supported on mechanical ventilation for acute respiratory failure in the PICU. Rather than seeking an elusive ideal drug, this unique nurse-led pilot study focuses on optimizing clinical decision making by: (a) multidisciplinary team education and consensus building; (b) multidisciplinary team identification of the patient's trajectory of illness and daily prescribing of a sedation goal; (c) a nurse-implemented sedation algorithm to guide titration of comfort medications; and(d)team feedback on clinical performance. This intervention models the most recent sedation clinical practice guideline published by the Society of Critical Care Medicine and addresses the only potentially manipulable factor influencing extubation failures rates in the Pediatric Intensive Care Unit.

The coordinating center, Children's Hospital Boston, developed, tested and currently uses the sedation algorithm as a standard of care. We will pilot the intervention in two separate previously selected PICUs that are matched on size and organization, academic affiliation and volume of patients supported on mechanical ventilation. One PICU will be randomized to receive early intervention while the other will first serve as a control, then will receive a delayed intervention.

The study design is a randomized controlled trial with delayed intervention in the control hospital. Because the intervention is an educational and organizational change directed at all PICU clinicians, the unit of randomization and analysis is the PICU. During the start-up phase, case report forms will be developed and a consensus meeting with all nurse and physician co-investigators will be conducted. The purpose of this consensus meeting will be to review the Children's Hospital Boston experience with the sedation algorithm and reach agreement on its application in the two PICUs. System nuances may impact protocol implementation and will require group discussion and multidisciplinary problem solving.

Study design includes baseline assessment of the organizational structure and comfort practices in both units. The PICU randomized to early intervention will then undergo training followed by implementation, a one-month respite, and post-data collection to evaluate the sustainability of the practice change. The PICU randomized to delayed intervention will start with pre-data collection, then undergo training followed by implementation. This design allows multiple comparisons; specifically, baseline to intervention/control, pre and post comparisons in both units, and sustainability in one unit.

Training will be multifaceted and will include all clinicians (physicians, nurses, clinical pharmacists and physicians-in-training) involved in the sedation management of intubated mechanically-ventilated patients. A multidisciplinary, cooperative approach is necessary to assure compliance and successful implementation of protocols. Training material will include discipline-specific lectures, informal discussions, video on sedation and opioid withdrawal scoring, bedside booklets, and physician order sheets. The research team will develop the supporting materials. Physician training will focus on sedation and opioid withdrawal scoring, identifying the patient's trajectory of illness, collaborating with nursing in prescribing the daily sedation goal, and completion of the standardized order template. Nursing content will likewise focus on sedation and opioid withdrawal scoring, trajectory analysis and collaboration, but also will include practical support on the daily "wake-up" test and titration of sedatives. Prior to the intervention phase, all physicians, physician-in-training, unit-based clinical pharmacist, charge nurses and full-time nursing staff will be required to document their understanding of the intervention by completion of a discipline-specific scenario-based self-assessment evaluation. Respiratory therapists will also require refresher instruction on extubation readiness testing and general information about sedation assessment and sedation algorithm.

During the implementation phase, daily multidisciplinary rounds will include identification of the patient's trajectory of illness and daily prescription of (a) sedation goal and (b) sedation parameters. Nurses will titrate the comfort medications as prescribed and perform a daily "wake up" test in patients during their stable phase who are not awake. During the implementation phase, a member of the research team will round separately on each patient to monitor for study compliance and offer staff support and re-training as necessary. This level of vigilance is necessary to identify aspects of the algorithm that are challenging to clinicians, and accurate reporting of protocol deviations requires an evaluation of the context of decision-making. This daily check will not continue in the early intervention arm when sustainability is evaluated. During the implementation phase, all sedation orders will be derived from standardized physician orders. This order template will serve two purposes: physician education and enhanced compliance with the algorithm

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated
* Pulmonary disease

Exclusion Criteria:

* Less than or equal to 2 weeks of age or 42 weeks corrected gestational age
* Greater than 18 years of age
* Intubated and mechanically ventilated for immediate post-operative care and stabilization
* Cyanotic heart disease with unrepaired or palliated right to left intracardiac shunt
* Critical airway (e.g. post laryngotracheal reconstruction)
* Ventilator dependent (including noninvasive) on PICU admission (chronic assisted ventilation)
* Neuromuscular respiratory failure
* Spinal cord injury above the lumbar region
* Managed by patient controlled analgesia (PCA)or epidural catheter
* Known allergy to any of the study medications (Morphine,Methadone, Midazolam, Lorazepam)
* Family/Medical team have decided not to provide full support(patient treatment considered futile)
* Previously enrolled into the current study or enrolled in any other sedation clinical trial concurrently or within the last 30 days

Ages: 2 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 245 (Actual)
Dates: Start 2004-02; Primary Completion 2006-07 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Duration of Mechanical Ventilation | 28 days

SECONDARY OUTCOMES:
Time to Recovery of Lung Injury | 28 days
Duration of Weaning from Mechanical Ventilation | 28 days
Occurrence of Adverse Events | 28 days
Total Exposure to Comfort Medications | 28 days
Occurrence of Iatrogenic Abstinence Syndrome | 28 days
PICU Length of Stay | 28 days
Barriers to Successful Implementation of the Intervention | 28 days
PICU costs | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Martha AQ Curley, RN PhD FAAN, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Curley MAQ, Gedeit RG, Dodson BL, Amling JK, Soetenga DJ, Corriveau CO, Asario LA, Wypij D; RESTORE Investigative Team. Methods in the design and implementation of the Randomized Evaluation of Sedation Titration for Respiratory Failure (RESTORE) clinical trial. Trials. 2018 Dec 17;19(1):687. doi: 10.1186/s13063-018-3075-8. PMID 30558653